CLINICAL TRIAL: NCT02994771
Title: A Phase I Open-Label Study to Assess the Safety, Tolerability and Preliminary Efficacy of Lymfactin® (AdAptVEGF-C Adenoviral Vector) in Combination With a Surgical Lymph Node Transfer for the Treatment of Patients With Secondary Lymphedema
Brief Title: A Phase I Study With Lymfactin® in the Treatment of Patients With Secondary Lymphedema
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Herantis Pharma Plc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL12001
Record Dates: First submitted 2016-11-10; First posted 2016-12-16 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Secondary Lymphedema
Keywords: Lymphedema, Breast cancer
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lymfactin® [1 x 10E10 vp] (Active Comparator): Lymfactin® [1 x 10E10 vp] will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Interventions: Drug: Lymfactin® [1 x 10E10 vp]
- Lymfactin® [1 x 10E11 vp] (Active Comparator): Lymfactin® [1 x 10E11 vp] will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Interventions: Drug: Lymfactin® [1 x 10E11 vp]

INTERVENTIONS:
Drug: Lymfactin® [1 x 10E10 vp] — Lymfactin® [1 x 10E10 vp] will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Other Names: LX-1101, AdAptVEGF-C Adenoviral Vector
  Arms: Lymfactin® [1 x 10E10 vp]
Drug: Lymfactin® [1 x 10E11 vp] — Lymfactin® [1 x 10E11 vp] will be administered as a single dose via perinodal injection in a volume of 2 mL.
  Other Names: LX-1101, AdAptVEGF-C Adenoviral Vector
  Arms: Lymfactin® [1 x 10E11 vp]

SUMMARY:
Indicated for the Treatment of Secondary Lymphedema Associated with the Treatment of Breast Cancer.

Primary objective is to evaluate the safety and tolerability of a single dose of Lymfactin® in patients with secondary lymphedema associated with the treatment of breast cancer.

DETAILED DESCRIPTION:
This is an open label, multi-center, uncontrolled first in human trial that uses a standard 3 + 3 dose escalation scheme. Lymfactin® will be administered as a single dose by ex vivo perinodal injection into the fat pad of a flap of tissue containing lymph nodes from the abdominal wall. This flap of tissue will then be surgically implanted into the axillary region of the affected arm. This treatment with Lymfactin® may be performed in conjunction with or without breast reconstruction surgery.

Up to two dose cohorts are planned to be included. Each dose of Lymfactin® will be administered as a single dose via perinodal injection in a volume of 2 mL:

* Cohort 1: Lymfactin® [1 x 10E10 vp]
* Cohort 2: Lymfactin® [1 x 10E11 vp]

Should the dose escalation go up to Cohort 2 with initiation of a subsequent Extension Cohort a total of 15 - 21 patients may be treated in this study.

ELIGIBILITY:
Inclusion criteria:

1. Female patients with secondary lymphedema associated with the treatment of breast cancer.
2. Patient who understands and voluntarily signs informed consent prior to any screening procedure.
3. 18 - 70 years of age.
4. BMI between 18 and 32 inclusive.
5. Female patients with secondary lymphedema in the arm associated with breast cancer who:

   1. Have undergone sentinel lymph node biopsies and/or lymph node resection in the axilla on the affected side of their breast cancer with initial N1 staging and lymph node metastasis in ≤ three lymph nodes.
   2. Require garment use as a compression treatment for the lymphedema in the affected arm.
   3. Have the volume of the affected arm at least 10% greater than the unaffected arm following 7 days after removal of the compression garments.
   4. Have the presence of pitting edema in the affected arm without compression garments.
6. No evidence of recurrent or active breast cancer at least 2 years and no more than 5 years after breast cancer surgery and/or the end of chemotherapy and/or radiotherapy (excluding endocrine and/or aromatase inhibitor treatment). PET CT scan of the chest and the abdomen within 45 days of treatment with Lymfactin® without signs of active breast cancer or any other malignancy.
7. Patient with the following laboratory values:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the institutional upper limit of normal (ULN)
   2. Bilirubin ≤ 1.5 mg/dL
   3. PT and PTT ≤ 1.5 times the ULN
   4. Serum creatinine ≤ 2 mg/dL
   5. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm³
   6. Platelet count ≥ 100,000/mm³
   7. Hemoglobin ≥ 10 g/dL
8. Willingness to comply with scheduled visits, laboratory assessments, and other study-related procedures due to the regulatory requirements related to gene based therapies.
9. Non-smoker or willing to stop smoking or using nicotine-containing products for at least 4 weeks prior to entry to study.
10. Negative urine pregnancy test (only patients with childbearing potential) at screening and use of adequate contraceptive measures from screening until 6 months after the study treatment administration:

    1. A patient with childbearing potential should be using a reliable contraception method: intrauterine device (hormonal or non-hormonal); oral combination pill or hormonal contraception patch; or two of the following: intra-vaginal hormonal ring, oral contraceptive containing progestin only, spermicidal foam, condom, sterilization of male sexual partner (surgical vasectomy).
    2. A patient with no current heterosexual relationship may be included according to the judgement of the Investigator.
    3. If the patient is surgically sterile or whose menopause occurred 2 years previously at the minimum, no contraception is required nor pregnancy test.

Exclusion criteria:

1. A patient who had an N2/N3 or a T4 stage breast cancer or an inflammatory breast cancer at the time of the original diagnosis.
2. A patient with evidence (clinical, laboratory, or imaging) or history of a neoplasm other than breast cancer (except basal cell carcinoma or cervical in situ carcinoma).
3. A patient known to be pregnant, lactating or having a positive or indeterminate pregnancy test.
4. Treatment with COX-2 inhibitors should be interrupted from one week prior until 2 weeks post surgery and treatment with Lymfactin®.
5. Previous treatment with, or participation in, trial of a gene therapy product.
6. Current participation or participation in the preceding two months, in any clinical study apart from a noninterventional study.
7. Current treatment with immunosuppressive drugs.
8. Current or history of drug, including nicotinecontaining products, or alcohol abuse.
9. Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
10. Allergy to any ingredients of the Lymfactin® solution for injection (glycerol, N-2-hydroxyethylpiperazine-N´-2-ethanesulfonic acid (HEPES), sodium hydroxide).
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, that would affect the patient's ability to follow study-related procedures, or that may interfere with the interpretation of study results and, in the Investigator's opinion, would make the patient inappropriate for entry into this study.
12. Doubtful availability, in the opinion of the Investigator, to complete the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Safety as measured by number of patients with treatment related adverse events and serious adverse events as assessed by CTCAE v4.0 | baseline to 1 year, yearly up to 5 years
  Adverse events and serious adverse events assessed by CTCAE v4.0 to evaluate the safety profile after administration of Lymfactin
CT scan of chest and abdomen | baseline, yearly up to 5 years
  Changes in the CT scan of chest and abdomen in order to detect malignancies
Biodistribution of Lymfactin in blood | 90 days
  Changes in Lymfactin genome copy number in blood
Formation of anti-Lymfactin antibodies | 6 months
  Changes in the anti-Lymfactin antibody titer in blood

SECONDARY OUTCOMES:
Measurement of the volume of the arms | baseline, 6, 12, 24 and 36 months
  Changes in the volume of the affected arm and comparison to the unaffected arm
Measurement of the lymphatic flow of the affected arm by quantitative lymphoscintigraphy (99Tc-nanocolloid clearance rate with calculation of transport index) | baseline, 12, 24 and 36 months
  Assessment of the changes in the lymphatic flow
Questionnaire according to the Lymphedema Quality of Life Inventory (LQOLI) | baseline, 6, 12, 24 and 36 months
  Assessment of changes in the quality of life using Lymphedema Quality of Life Inventory (LQOLI) in which patients assess how their lymphedema is affecting the activities of daily living. LQOLI consists of three dimensions: Physical, psychosocial and practical, which are reported separately as the mean score of each dimension. Each dimension of the LQOLI is scored from 0 to 3, where score 0 means "no impact", 1 means "a little bit impact", 2 means "somewhat impact", and 3 means "significant impact" on the quality of life of the patient, the smaller score thus being the better.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Saarikko, MD, PhD, Principal Investigator — HUCH
Locations (3):
- Finland (3):
  - Toeoeloe Hospital, Department of Plastic Surgery, Helsinki
  - Tampere University Hospital, Department of Plastic Surgery, Tampere
  - Turku University Hospital, Department of Plastic Surgery, Turku

IPD SHARING:
Plan to Share IPD: No